CLINICAL TRIAL: NCT04220866
Title: A Phase 2 Study in First Line Metastatic or Unresectable, Recurrent Head and Neck Squamous Cell Carcinoma to Evaluate Intratumoral MK-1454 in Combination With IV Pembrolizumab vs IV Pembrolizumab Monotherapy
Brief Title: Study of Intratumoral (IT) Ulevostinag (MK-1454) in Combination With Intravenous (IV) Pembrolizumab (MK-3475) Compared to IV Pembrolizumab Alone as the First Line Treatment of Metastatic or Unresectable, Recurrent Head and Neck Squamous Cell Carcinoma (HNSCC) (MK-1454-002)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1454-002; MK-1454-002 (Other: Merck); 2019-003060-42 (EudraCT Number)
Record Dates: First submitted 2020-01-06; First posted 2020-01-07 (Actual); Results first posted 2023-10-27 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Head and Neck Squamous Cell Carcinoma (HNSCC)
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1); intratumoral (IT); metastatic; unresectable; recurrent; ulevostinag; pembrolizumab
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Parkinson Disease 4, Autosomal Dominant Lewy Body; Neoplasm Metastasis; Recurrence | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ulevostinag+Pembrolizumab (Experimental): Participants receive ulevostinag 540 ug via intratumoral (IT) injection on Day 1 of every week for two 3-week cycles (Cycles 1-2), then on Day 1 of each 3-week cycle for up 33 cycles (Cycles 3-35), for a total of 35 cycles PLUS pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 35 cycles. The total duration of treatment is up to approximately 2 years.
  Interventions: Drug: Ulevostinag; Biological: Pembrolizumab
- Pembrolizumab (Active Comparator): Participants receive pembrolizumab 200 mg via IV infusion on Day 1 of each 3-week cycle for up to 35 cycles. The total duration of treatment is up to approximately 2 years.
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Drug: Ulevostinag — IT injection
  Other Names: MK-1454
  Arms: Ulevostinag+Pembrolizumab
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®

SUMMARY:
The purpose of this study is to assess the efficacy and safety of intratumoral (IT) ulevostinag PLUS pembrolizumab (MK-3475) compared to pembrolizumab alone as a first line treatment of adults with metastatic or unresectable, recurrent head and neck squamous cell carcinoma (HNSCC).

The primary study hypotheses are that IT ulevostinag in combination with pembrolizumab results in a superior Objective Response Rate (ORR), per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1), compared to pembrolizumab alone:

1. In participants with a tumor that has a programmed cell death-ligand 1 (PD-L1) Combined Positive Scoring (CPS) ≥ 1, and
2. In participants with a tumor that has a PD-L1 CPS ≥ 20.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically or cytologically confirmed diagnosis of metastatic or unresectable, recurrent head and neck squamous cell carcinoma (HNSCC) that is considered incurable by local therapies
* Has not had prior systemic therapy administered in the recurrent or metastatic setting
* Has tumor PD-L1 expression of CPS ≥1. Tumor tissue must be provided for PD-L1 biomarker analysis
* Has measurable disease per RECIST 1.1, as assessed by BICR
* Has at least 1 measurable lesion which is amenable to injection
* Has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Demonstrates adequate organ function within 7 days prior to treatment initiation
* Male participants of reproductive potential must agree to refrain from donating sperm and use a male condom plus partner use of an additional contraceptive method during sexual contact with females of childbearing potential during the intervention period with ulevostinag and for at least 120 days after the last dose of ulevostinag
* Female participants of childbearing potential who are not pregnant or breastfeeding must be willing to use a highly effective method of birth control or be surgically sterile or abstain from heterosexual activity during the intervention period and for at least 120 days after the last dose of study intervention, and agree not to donate eggs (ova, oocytes) to others or freeze/store for personal use
* Human immunodeficiency virus (HIV)-infected participants must meet these additional criteria:

  1. Has HIV-1 infection documented by using any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry (Day 1)
  2. Has well-controlled HIV on anti-retroviral therapy (ART)

Exclusion Criteria:

* Has disease that is suitable for local therapy administered with curative intent
* Has progressive disease (PD) within 6 months of completion of curatively intended systemic treatment for locoregionally advanced HNSCC
* Has had chemotherapy or biological cancer therapy in the recurrent or metastatic setting for the treatment of HNSCC
* Has had radiation therapy (or other non-systemic therapy) within 2 weeks prior to randomization or participant has not fully recovered from adverse events (AEs) due to a previously administered treatment
* Is expected to require any other form of antineoplastic therapy while on study
* Has a history of a second malignancy, unless potentially curative treatment has been completed, with no evidence of malignancy for at least 2 years
* Has clinically active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has an active autoimmune disease that has required systemic treatment in the past 2 years
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment
* Has had an allogenic tissue/solid organ transplant
* Has a history of vasculitis
* Has a history of interstitial lung disease
* Has an active infection requiring systemic therapy
* Has a known history of active tuberculosis (TB; Bacillus tuberculosis)
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Has had a severe hypersensitivity reaction to treatment a monoclonal antibody/components of the study treatment
* Has known Hepatitis B virus or Hepatitis C virus infections
* Has received prior therapy with an anti-programmed cell death 1 (anti-PD-1), anti-programmed cell death-ligand 1 (anti-PD-L1), or anti-programmed cell death-ligand 2 (anti-PD-L2) agent or if the participant has previously participated in Merck Sharp & Dohme (MSD) MK-3475 clinical trials
* HIV infected participant who has had an HIV-related opportunistic infection within 6 months
* HIV infected participants who have a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Is pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment
* Has not fully recovered from any effects of major surgery without significant detectable infection
* Has a history of re-irradiation for HNSCC at the projected injection site in the head and neck
* Has received a live-virus vaccine within 30 days of planned study treatment start
* Has been treated with a stimulator of interferon genes (STING) agonist (e.g. ulevostinag, ADU-S100)
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy, or used an investigational device, any of which occurred within 4 weeks of the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (34):
- United States (6):
  - UCLA Hematology & Oncology ( Site 0005), Los Angeles, California
  - University of California at San Francisco ( Site 0006), San Francisco, California
  - Henry Ford Hospital ( Site 0012), Detroit, Michigan
  - Washington University ( Site 0021), St Louis, Missouri
  - Sanford Cancer Center Oncology Clinic ( Site 0014), Sioux Falls, South Dakota
  - Huntsman Cancer Institute ( Site 0004), Salt Lake City, Utah
- Australia (3):
  - Chris OBrien Lifehouse ( Site 0040), Camperdown, New South Wales
  - Calvary Central Districts Hospital ( Site 0042), Elizabeth Vale, South Australia
  - Monash Health-Monash Medical Centre ( Site 0041), Clayton, Victoria
- Austria (3):
  - Ordensklinikum Linz Gmbh - Barmherzige Schwestern ( Site 0051), Linz, Upper Austria
  - Allgemeines Krankenhaus der Stadt Wien ( Site 0049), Vienna/Wien, Vienna
  - SCRI-CCCIT GesmbH ( Site 0050), Salzburg
- Brazil (4):
  - Centro Regional Integrado de Oncologia ( Site 0062), Fortaleza, Ceará
  - Hospital de Caridade de Ijui ( Site 0061), Ijuí, Rio Grande do Sul
  - Instituto do Cancer do Estado de Sao Paulo - ICESP ( Site 0058), São Paulo
  - Real e Benemerita Associacao Portuguesa de Beneficencia ( Site 0064), São Paulo
- France (5):
  - Centre Antoine Lacassagne ( Site 0070), Nice, Alpes-Maritimes
  - Centre Leon Berard ( Site 0072), Lyon, Auvergne
  - IUCT - Oncopole ( Site 0069), Toulouse, Haute-Garonne
  - Centre Oscar Lambret ( Site 0071), Lille, Nord
  - Gustave Roussy ( Site 0068), Villejuif, Val-de-Marne
- Israel (3):
  - Chaim Sheba Medical Center ( Site 0076), Ramat Gan, Tel Aviv
  - Rambam Medical Center ( Site 0077), Haifa
  - Hadassah Medical Center. Ein Kerem ( Site 0078), Jerusalem
- Norway (2):
  - Haukeland Universitetssykehus, Klinisk forskningspost voksne ( Site 0086), Bergen, Hordaland
  - Oslo Universitetssykehus Radiumhospitalet ( Site 0085), Oslo
- South Korea (2):
  - Severance Hospital ( Site 0103), Seoul
  - Asan Medical Center ( Site 0104), Seoul
- Spain (4):
  - H.U. Vall de Hebron ( Site 0112), Barcelona
  - Hospital Clinico de Barcelona ( Site 0116), Barcelona
  - Hospital Universitario Ramon y Cajal ( Site 0115), Madrid
  - Hospital Universitario Virgen de la Victoria ( Site 0114), Málaga
- United Kingdom (2):
  - Royal Marsden NHS Foundation Trust ( Site 0031), London, London, City of
  - Royal Marsden Hospital Sutton-Surrey ( Site 0032), Sutton, Surrey

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Harrington KJ, Champiat S, Brody JD, Cho BC, Romano E, Golan T, Hyngstrom JR, Strauss J, Oh DY, Popovtzer A, Gomez-Roca C, Perets R, Kim SB, Wong DJ, Powell SF, Khilnani A, Jemielita T, Zhao Q, Zhao R, Ingham M. Phase I and II Clinical Studies of the STING Agonist Ulevostinag with and without Pembrolizumab in Participants with Advanced or Metastatic Solid Tumors or Lymphomas. Clin Cancer Res. 2025 Aug 14;31(16):3400-3411. doi: 10.1158/1078-0432.CCR-24-3630. PMID 40499147
- [Derived] McIntosh JA, Liu Z, Andresen BM, Marzijarani NS, Moore JC, Marshall NM, Borra-Garske M, Obligacion JV, Fier PS, Peng F, Forstater JH, Winston MS, An C, Chang W, Lim J, Huffman MA, Miller SP, Tsay FR, Altman MD, Lesburg CA, Steinhuebel D, Trotter BW, Cumming JN, Northrup A, Bu X, Mann BF, Biba M, Hiraga K, Murphy GS, Kolev JN, Makarewicz A, Pan W, Farasat I, Bade RS, Stone K, Duan D, Alvizo O, Adpressa D, Guetschow E, Hoyt E, Regalado EL, Castro S, Rivera N, Smith JP, Wang F, Crespo A, Verma D, Axnanda S, Dance ZEX, Devine PN, Tschaen D, Canada KA, Bulger PG, Sherry BD, Truppo MD, Ruck RT, Campeau LC, Bennett DJ, Humphrey GR, Campos KR, Maddess ML. A kinase-cGAS cascade to synthesize a therapeutic STING activator. Nature. 2022 Mar;603(7901):439-444. doi: 10.1038/s41586-022-04422-9. Epub 2022 Mar 16. PMID 35296845
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults with a confirmed diagnosis of metastatic or unresectable, recurrent head and neck squamous cell carcinoma (HNSCC) with a tumor programmed cell death-1 ligand 1 (PD-L1) immunohistochemistry (IHC) combined positive scoring (CPS) ≥1 and had at least 1 measurable lesion that was amenable to intratumor (IT) injection were enrolled in this study.
Groups:
- Ulevostinag + Pembrolizumab: Participants received ulevostinag 540 ug via intratumoral (IT) injection on Day 1 of every week for two 3-week cycles (Cycles 1-2), then on Day 1 of each 3-week cycle for up 33 cycles (Cycles 3-35), for a total of 35 cycles PLUS pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 35 cycles. The total duration of treatment was up to approximately 2 years.
- Pembrolizumab: Participants received pembrolizumab 200 mg via IV infusion on Day 1 of each 3-week cycle for up to 35 cycles. The total duration of treatment is up to approximately 2 years.
Period: Overall Study
Arm/Group | Ulevostinag + Pembrolizumab | Pembrolizumab
Started (Randomized) | 8 | 10
Completed | 0 | 0
Not Completed | 8 | 10
Not completed — Death | 4 | 5
Not completed — Participation at the site terminated By Sponsor | 2 | 0
Not completed — Participation in the study terminated By Sponsor | 2 | 4
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Ulevostinag + Pembrolizumab: Participants received ulevostinag 540 ug via IT injection on Day 1 of every week for two 3-week cycles (Cycles 1-2), then on Day 1 of each 3-week cycle for up 33 cycles (Cycles 3-35), for a total of 35 cycles PLUS pembrolizumab 200 mg via intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 35 cycles. The total duration of treatment was up to approximately 2 years.
- Total: Total of all reporting groups
Arm/Group | Ulevostinag + Pembrolizumab | Pembrolizumab | Total
Number analyzed (Participants) | 8 | 10 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.3 (9.8) | 59.8 (9.8) | 62.2 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 8 | 9 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 10 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 9 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: ORR was defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. ORR was assessed by blinded independent central review (BICR), and the 95% confidence interval (CI) was based on the exact method for binomial data.
Time Frame: Up to 913.0 days
Population: All randomized participants based on the treatment arm to which they were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ulevostinag + Pembrolizumab | Pembrolizumab
Number analyzed (Participants) | 8 | 10
Percentage of participants | 50.0 [15.7 to 84.3] | 10.0 [0.3 to 44.5]

2. Secondary Outcome: Progression-free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) or death from any cause, whichever occurs first. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered PD. PFS was assessed by BICR and was based on the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to 913.0 days
Population: All randomized participants based on the treatment arm to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ulevostinag + Pembrolizumab | Pembrolizumab
Number analyzed (Participants) | 8 | 10
Months | 6.4 [1.0 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 1.5 [0.5 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event.

3. Secondary Outcome: Duration of Response (DOR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: DOR was defined as the time from the first documented evidence of a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 until Progressive Disease (PD) or death due to any cause, whichever occurs first, in participants demonstrating a CR or PR. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR was based on the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to 913.0 days
Population: All randomized participants based on the treatment arm to which they were randomized.
Measure: Median (Full Range); unit: Months
Arm/Group | Ulevostinag + Pembrolizumab | Pembrolizumab
Number analyzed (Participants) | 8 | 10
Months | NA [4.2 to 30.4] — NA = Median not reached at time of data cut-off due to insufficient number of responding participants with relapse. | NA [1.4 to 1.4] — NA = Median, not reached at time of data cut-off due to insufficient number of responding participants with relapse.

4. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization to the date of death from any cause, and is based on the product-limit (Kaplan-Meier) method for censored data.
Time Frame: Up to 913.0 days
Population: All randomized participants based on the treatment arm to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ulevostinag + Pembrolizumab | Pembrolizumab
Number analyzed (Participants) | 8 | 10
Months | NA [1.0 to NA] — NA = Median and upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 11.1 [0.8 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event.

5. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Time Frame: Up to 913.0 days
Population: All randomized participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ulevostinag + Pembrolizumab | Pembrolizumab
Number analyzed (Participants) | 8 | 10
Participants | 8 | 10

6. Secondary Outcome: Number of Participants Discontinuing Study Treatment Due to an AE
Description: as for outcome 5
Time Frame: Up to approximately 715.0 days
Population: All randomized participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ulevostinag + Pembrolizumab | Pembrolizumab
Number analyzed (Participants) | 8 | 10
Participants | 3 | 2

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs): from first treatment up to 913.0 days. All Cause Mortality (ACM): from randomization up to 913.0 days.:
Description: The population analyzed for ACM consisted of all randomized participants. The population for AEs consisted of all randomized participants who received at least1 dose of study treatment. Per protocol disease progression of cancer was not considered an AE unless related to study drug. Therefore the following AE preferred terms not related to the drug were excluded: Neoplasm progression, Malignant neoplasm progression and Disease progression.
Arm/Group | Ulevostinag + Pembrolizumab | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 4/8 | 5/10
Serious Adverse Events (participants affected / at risk) | 5/8 | 4/10
Other Adverse Events (participants affected / at risk) | 8/8 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ulevostinag + Pembrolizumab (N=8) | Pembrolizumab (N=10)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Injection site ulcer (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Injection related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carotid artery aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ulevostinag + Pembrolizumab (N=8) | Pembrolizumab (N=10)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hyperacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Palatal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (4) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1)
Axillary pain (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 2 (5) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 1 (2) | 0 (0)
Injection site necrosis (General disorders) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 4 (6) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 4 (10) | 0 (0)
Swelling (General disorders) | 1 (1) | 0 (0)
Swelling face (General disorders) | 1 (2) | 0 (0)
Bacterial disease carrier (Infections and infestations) | 1 (1) | 0 (0)
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1)
Candida infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (2) | 0 (0)
Pyuria (Infections and infestations) | 1 (1) | 0 (0)
Relapsing fever (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Tongue fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stoma site discharge (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
Tri-iodothyronine free increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neoplasm swelling (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Skin neoplasm bleeding (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour inflammation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anosmia (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nasal cavity mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Sensitive skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT04220866/Prot_SAP_000.pdf